CLINICAL TRIAL: NCT01845259
Title: Does a GLP-1 Receptor Agonist Change Glucose Tolerance in Antipsychotic-treated Patients? A Randomized, Double-blinded, Placebo-controlled Clinical Trial
Brief Title: Does a GLP-1 Receptor Agonist Change Glucose Tolerance in Antipsychotic-treated Patients?
Acronym: GREAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); University of Cambridge (Other)
Responsible Party: Principal Investigator, Anders Fink-Jensen, MD, DMSci, Professor, MD, DMSci, Psychiatric Centre Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLP-1 antipsychotics; 2013-000121-31 (EudraCT Number); U1111-1128-3404 (Registry Identifier: UTN-number)
Record Dates: First submitted 2013-04-14; First posted 2013-05-03 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Impaired Glucose Tolerance Associated With Drugs
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): Once a day 1,8 mg subcutaneous injection for 16 weeks
  Interventions: Drug: Liraglutide
- Liraglutide placebo (Placebo Comparator): Once a day 1,8 mg subcutaneous injection for 16 weeks
  Interventions: Drug: Liraglutide Placebo

INTERVENTIONS:
Drug: Liraglutide — Once a day 1,8 mg subcutaneous injection for 16 weeks
  Other Names: Victoza; GLP-1 agonist
  Arms: Liraglutide
Drug: Liraglutide Placebo — Once a day 1,8 mg subcutaneous injection for 16 weeks
  Other Names: Placebo
  Arms: Liraglutide placebo

SUMMARY:
Metabolic disturbances, obesity and life-shortening cardiovascular morbidity are major clinical problems among antipsychotic-treated patients. Especially two of the most efficacious antipsychotics, clozapine and olanzapine, cause weight gain and metabolic disturbances and can rarely be replaced by other drugs due to the effectiveness of the compounds. Glucagon-like peptide 1 (GLP-1) has improved glycemic control among patients with type 2 diabetes. The study will investigate whether the beneficial effects of GLP-1 analogues on glycemic control in type 2 diabetic patients, can be extended to a population of non-diabetic, dysglycemic psychiatric patients, receiving antipsychotic medical treatment.

DETAILED DESCRIPTION:
Statistical analyses:

Power calculation:

A sample size of 96 participants (48 in each group) was estimated, with two-sided t-testing, an α of 5% and a power of 90%. The power calculation was based on the primary outcome measurement: Change in glucose tolerance. The glucose tolerance was estimated by the total Area Under the Curve (AUC) following a 4-hour 75-g. Oral Glucose Tolerance Test (OGTT). The expected mean total AUC for the plasma glucose excursion following a 4-hour 75-g. OGTT was estimated as 1695 (SD 158) and 1800 (SD 158) after 16 weeks of treatment for the liraglutide and liraglutide placebo group, respectively. The difference in total AUC was based on unpublished data in individuals with and without Impaired Glucose Tolerance (IGT) following a 4-hour 75-g. OGTT at baseline from the study: "The Impact of Liraglutide on Glucose Tolerance and the Risk of Type 2 Diabetes in Women With Previous Pregnancy-induced Diabetes".(1)

Procedure:

All analyses will be carried out with the treatment groups still blinded and labeled as "treatment group A" and "treatment group B". Before dividing participants into group A and group B, the statistical plan was completed and uploaded on clinicaltrials.gov, and the data set was locked. The final unblinding of treatment groups (liraglutide or liraglutide placebo), will not be carried out until all statistical analyses are performed. All analyses will be performed using SAS 9.4, with α set at 0.05 and two-sided testing.

All efficacy analyses will be performed using a modified intention-to-treat principle. All participants who were randomized, received at least one dose of the trial compound (liraglutide or liraglutide placebo) and who had at least one assessment after baseline will be included in the efficacy analyses. All safety analyses will be performed in the intent-to-treat sample that includes all participants, who were randomized and received at least one dose of the trial compound (liraglutide or liraglutide placebo).

Primary endpoint:

The primary endpoint is the change in glucose tolerance following a 4-hour 75-g. OGTT from week 0 to week 16. During the 4-hour 75-g. OGTT, blood was sampled at fixed time points: -15, -10, 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, and 240 minutes. An analysis of covariance (ANCOVA) will be use to analyze change in glucose tolerance from week 0 to week 16 using mixed model analyses for the plasma glucose levels for the liraglutide and the liraglutide placebo group, respectively. In case of relevant baseline differences between the two groups, demographic, illness or treatment parameters will be included in the model as fixed effects together with the baseline value of the OGTTs as a covariate.

Secondary endpoints:

Blood was also sampled for analyses of C-peptide, glucagon and incretin hormones in response to the glucose load at the same fixed time points during the OGTT. Change in secretion of C-peptide, glucagon and incretin hormones from week 0 to week 16 will also be evaluated using mixed model ANCOVA analyses for the liraglutide and liraglutide placebo group, respectively. In case of relevant baseline differences between the two groups, demographic, illness or treatment parameters will be included in the model as fixed effects together with the baseline value of the relevant variable as a covariate.

Most secondary endpoints were repeated every 4 weeks. Few secondary endpoints were only repeated at week 0 and 16. For all repeated measurements a mixed model ANCOVA analyses will be use to analyze mean change in continuous outcomes from week 0 to week 16 for the liraglutide and the liraglutide placebo group, respectively. In case of relevant baseline differences between the two groups, demographic, illness or treatment parameters will be included in the model as fixed effects together with the baseline value of the relevant variable as a covariate. Change in categorical outcomes from week 0 to week 16 will be analyzed using mixed model logistic regression with the same fixed effects and covariates as described for the continuous outcomes.

For secondary endpoints without repeated measurements, missing data imputations will be made using Multiple Imputation of Chained Equations (MICE).

For continuous outcomes without repeated measurements, outcomes will be analyzed using ANCOVA to detect differences between the liraglutide and the liraglutide placebo group. In the model baseline demographic, illness or treatment parameters will be included. Categorical outcomes without repeated measurements will be analyzed using a multiple mixed effect logistic regression analysis model, where baseline demographic, illness or treatment parameters will be included.

Subgroup and sensitivity analyses:

Subgroup and sensitivity analyses will be performed to assess the robustness of the primary analyses. These analyses will be performed using regression analysis for continuous outcomes and logistic regression for categorical outcomes. The analyses will consider clinically or mechanistically relevant baseline and intra-treatment variables, including:

* Gender
* Smoking
* Antipsychotics (clozapine vs olanzapine; monopharmacy vs polypharmacy with other antipsychotic medications)
* Lipid profile
* Liver function
* Different groups of dysglycaemia:

  1. HbA1c: 43 mmol/mol ≤ HbA1c ≤ 47 mmol/mol, vs
  2. Impaired fasting glucose (IFG): Fasting plasma glucose (FPG): 6.1 mmol/l ≤ FPG ≤ 6.9 mmol/l and HbA1c < 48 mmol/mol, vs
  3. Impaired glucose tolerance (IGT): two-hour plasma glucose after 75-g oral glucose tolerance test >7.8 mmol/l with a FPG < 7.0 mmol/l and HbA1c < 48 mmol/mol
* IGT < 11 mmol/l vs IGT >11 mmol/l
* Liraglutide treatment (1.2 mg vs 1.8 mg liraglutide)
* Weight
* Add-on psychotropic drugs/classes (antidepressants, anxiolytics etc. vs no add-on)
* Antihypertensive treatment vs no antihypertensive treatment
* Lipid lowering treatment vs no lipid lowering treatment
* Changes in antipsychotic medication (> 20 % change in dose vs < 20 % change in dose vs no changes in dose for clozapine or olanzapine, respectively)
* Inhalation steroid vs no inhalation steroid
* Body composition
* Insulin resistance
* Beta-cell function
* Incretin hormones
* Psychopathologic rating scales
* Alcohol consumption
* Length of disease
* Diagnosis (schizophrenia vs schizotypal disorder vs paranoid psychosis)
* Side effects
* Serious adverse events

Reference List

1. Foghsgaard S, Vedtofte L, Mathiesen ER et al. The effect of a glucagon-like peptide-1 receptor agonist on glucose tolerance in women with previous gestational diabetes mellitus: protocol for an investigator-initiated, randomised, placebo-controlled, double-blinded, parallel intervention trial. BMJ Open 2013;3(10):e003834.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Diagnosed with schizophrenia, schizotypal disorder or paranoid psychosis according to the criteria of ICD10 (International Classification of Diseases, World Health Organization) or the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, the American Psychiatric Association)
* and on stable antipsychotic treatment with either clozapine or olanzapine for at least 6 months (without dose change for at least 30 days)
* Stable co-medications for at least 30 days.
* Age ≥18 years and ≤65 years
* Stable weight (defined as less than 5% change in weight over the last 3 month before inclusion)
* BMI ≥27 kg/m2
* Dysglycaemia (IFG, i.e. fasting plasma glucose level from 6.1 mmol/L to 6.9 mmol/L or IGT, i.e. two-hour glucose levels > 7.8 mmol/L on the 75-g oral glucose tolerance test with a fasting plasma glucose of less than 7.0 mmol/L and HbA1c < 48 mmol/mol or HbA1c: 43 mmol/mol ≤ HbA1c ≤ 47 mmol/mol)

Exclusion Criteria:

* Compulsory treatment
* Females of child bearing potential who are pregnant, breast-feeding or have intention of becoming pregnant or are not using adequate contraceptive measures
* Subjects treated with corticosteroids or other hormone therapy (except estrogens)
* Any active substance abuse or dependence for the past 6 months (except for nicotine)
* Impaired hepatic function (liver transaminases >2 times upper normal limit)
* Impaired renal function (se-creatinine >150 μM and/or macroalbuminuria)
* Impaired pancreatic function (acute or chronic pancreatitis and/or amylase >2 times upper normal limit)
* Cardiac problems defined as decompensated heart failure (NYHA class III or IV), unstable angina pectoris and/or myocardial infarction within the last 12 months
* Uncontrolled hypertension (systolic blood pressure >180 mmHg, diastolic blood pressure >100 mmHg)
* Any condition that the investigator feels would interfere with trial participation
* Receiving any investigational drug within the last 3 months
* Use of weight-lowering pharmacotherapy within the preceding 3 month
* Type 1 or 2 diabetes with HbA1c > 6.5%

Also a group of healthy controls (n=10) will have the baseline examinations done. The healthy controls will be matched to our participants in regards to gender, BMI and age. The same inclusion and exclusion criteria will apply for these controls, except these participants are not allowed to have known psychiatric illness, receive anti-psychotic medications, or have a family history of type 2 diabetes (2 generations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance | Baseline - 16 weeks
  Change in Glucose tolerance (measured by area under the curve (AUC) for plasma glucose (PG) excursion following a 4-hour 75 g Oral Glucose Tolerance Test (OGTT))

SECONDARY OUTCOMES:
Dysglycaemia | Baseline - 16 weeks
  Change in dysglycaemia (Impaired Fasting Glucose (IFG), Impaired Glucose Tolerance (IGT), combined IFG/IGT or diabetes)
Body weight | Every 4 weeks from baseline - 16 weeks
Secretion of incretin hormons, insulin sensitivity and beta cell function | Baseline - 16 weeks
  Evaluated by Homeostatic Model of Assessment (HOMA)
Body composition | Baseline - 16 weeks
  Dual energy x-ray absorptiometry (DEXA)-scan
Lipid profile and liver function | Every 4 weeks from baseline - 16 weeks
  Blood sample
Psychopathology | Baseline - 16 weeks
  Schizophrenia Quality of Life Scale (SQLS), Clinical Global Impression-Severity (CGI-S), Clinical Global Impression-Improvement (CGI-I), Global Assessment of Function (GAF)
Waist circumference | Every 4 weeks from baseline - 16 weeks
Blood pressure | Every 4 weeks from baseline - 16 weeks

OTHER OUTCOMES:
Alcohol use | Every 4 weeks from baseline - 16 weeks
  AUDIT (Alcohol Use Disorder Identification Test)
Changes i dietary and exercise records | Every 4 weeks from baseline - 16 weeks
Proteomic fingerprinting | Every 4 weeks from baseline - 16 weeks
  We wish to identify baseline imbalances among our participants with proteomic fingerprinting. Furthermore, we will test the dysglycemic and metabolic disturbances in patients treated for 16 weeks with liraglutide or placebo. We wish to investigate, whether treatment with liraglutide possible could rebalance some of the metabolic, immune and hormonal disturbances, we expect to find at baseline.
Long term follow-up 52 weeks after end of participation | 52 weeks after 16 weeks of liraglutide/placebo-treatment
  The follow-up 52 weeks after end of participation will include:
  • Medical history: Changes in antipsychotic medication Changes in other medications Changes in diet and exercise habits Changes in smoking Diagnosed with diabetes or other diseases
  * Blood sampling
  * Blood pressure
  * Weight
  * Height
  * Waist circumference
  * Alcohol Use Disorder Identification Test (AUDIT)
  * Schizophrenia Quality of Life Scale (SQLS)
  * Clinical Global Impression-Severity and Improvement (CGI-S+I)
  * Global Assessment of Function (GAF)
Baseline comparisons with healthy controls (non-psychiatric, non-diabetic) | Baseline examination
  In order to identify risk factors for diabetes development in individuals on antipsychotic medications, the baseline examinations will be performed on a group of healthy controls without psychiatric illnes or pre-diabetes (n=10). The healthy controls will be matched to our participants in regards to gender, age and BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fink-Jensen, MD, DMSci, Principal Investigator — Psychiatric Centre Rigshospitalet; Tina Vilsbøll, MD, DMSci, Principal Investigator — Diabetes Research Division, Gentofte
Locations (1):
- Psychiatric Centre Rigshospitalet, Copenhagen, København Ø, Denmark

REFERENCES:
- [Derived] Larsen JR, Vedtofte L, Jakobsen MSL, Jespersen HR, Jakobsen MI, Svensson CK, Koyuncu K, Schjerning O, Oturai PS, Kjaer A, Nielsen J, Holst JJ, Ekstrom CT, Correll CU, Vilsboll T, Fink-Jensen A. Effect of Liraglutide Treatment on Prediabetes and Overweight or Obesity in Clozapine- or Olanzapine-Treated Patients With Schizophrenia Spectrum Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jul 1;74(7):719-728. doi: 10.1001/jamapsychiatry.2017.1220. PMID 28601891
- [Derived] Sharma AN, Ligade SS, Sharma JN, Shukla P, Elased KM, Lucot JB. GLP-1 receptor agonist liraglutide reverses long-term atypical antipsychotic treatment associated behavioral depression and metabolic abnormalities in rats. Metab Brain Dis. 2015 Apr;30(2):519-27. doi: 10.1007/s11011-014-9591-7. Epub 2014 Jul 15. PMID 25023888
- [Derived] Larsen JR, Vedtofte L, Holst JJ, Oturai P, Kjaer A, Correll CU, Vilsboll T, Fink-Jensen A. Does a GLP-1 receptor agonist change glucose tolerance in patients treated with antipsychotic medications? Design of a randomised, double-blinded, placebo-controlled clinical trial. BMJ Open. 2014 Mar 25;4(3):e004227. doi: 10.1136/bmjopen-2013-004227. PMID 24667381